CLINICAL TRIAL: NCT00792571
Title: An Open-Label Extension of BPS-MR-PAH-201 in Pulmonary Arterial Hypertension (PAH) Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lung Biotechnology PBC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPS-MR-PAH-202
Record Dates: First submitted 2008-11-14; First posted 2008-11-18 (Estimated); Results first posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- B.I.D (Experimental): Beraprost Sodium Modified Release Tablets, 60mcg, b.i.d (twice a day dosing)
  Interventions: Drug: Beraprost Sodium Modified Release
- Q.I.D (Experimental): Beraprost Sodium Modified Release Tablets, 60mcg, q.i.d (four times a day dosing)
  Interventions: Drug: Beraprost Sodium Modified Release

INTERVENTIONS:
Drug: Beraprost Sodium Modified Release
  Other Names: BPS-MR Tablets, 60 mcg; Beraprost Sodium Modified Release Tablet, 60 mcg

SUMMARY:
This is an open-label extension study for patients who participated in the BPS-MR-PAH-201 study.

DETAILED DESCRIPTION:
This is an open-label study for patients who participated in the BPS-MR-PAH-201 study and have volunteered to continue treatment for PAH with BPS-MR tablets. Each patient will return to the clinic following enrollment in the study at 3, 6, and 12 months, and annually thereafter for assessment.

Currently enrolled patients may be invited to participate in an optional four times daily (QID) dosing substudy of BPS-MR with total daily dose of BPS-MR achieved previously in the main study. Patients will return to the clinic for baseline visit, week 12, and then will follow the visit schedule provided to them in BPS-MR-PAH-202 main study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who remained on study drug and completed all assessments during the Treatment Phase of Study BPS-MR-PAH-201 are eligible for this study.
* Female patients must either be physiologically incapable of childbearing or be practicing an acceptable method of birth control (e.g. approved hormonal contraceptive, barrier method, such as condom or diaphragm, used with a spermicide, or an intrauterine device).

Exclusion Criteria:

* Patients who discontinued study drug during the previous study (BPS-MR-PAH-201) for any reason (e.g. treatment related adverse events) are not eligible for entry into this study.
* Patients who are pregnant or lactating are excluded from participation in the open-label extension.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-02-28 (Actual); Primary Completion 2013-11-30 (Actual); Study Completion 2013-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Smart, Study Director — Study Sponsor
Locations (6):
- United States (3):
  - Harbor-UCLA Medical Center, Torrance, California
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UTSW Medical Center Dallas, Dallas, Texas
- Belgium (2):
  - Universite Libre de Bruxelles, Brussels
  - Gastuisberg University Hospital, Leuven
- Mater Misericordiae University Hospital Ltd., Dublin, Ireland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with pulmonary artery hypertension (PAH) who had completed lead in study BPS-MR-PAH-201 were enrolled in this study
Pre-assignment Details: A Protocol Amendment was to include an optional arm investigating Beraprost Sodium Modified Release Tablets administered four times daily (QID), however, no participants were enrolled into this arm.
Groups:
- Beraprost Sodium: Beraprost Sodium Modified Release Tablets, 60mcg, b.i.d (twice a day dosing)
Period: Overall Study
Arm/Group | Beraprost Sodium
Started | 18
Completed | 8
Not Completed | 10
Not completed — Death | 1
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 1
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (13.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Six-Minute Walk Distance [Mean (Standard Deviation); unit: meters] — A 6 minute walk test (6MWT) was conducted that measured how far a participant could walk in 6 continous minutes. Participants were instructed to walk as far as possible in 6 minutes, and were allowed to slow down and take breaks as needed due to symptoms.
  meters | 419.5 (73.1)
Borg Dyspnea Score [Mean (Standard Deviation); unit: score on a scale] — The Modified Borg scale was an 11 point scale with a score range of 0-10, where 0 indicated no breathlessness at all and 10 indicated maximum breathlessness.
  score on a scale | 3.4 (2.44)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting at Least One Treatment-Emergent Adverse Event (TEAE)
Description: A treatment-emergent adverse event (TEAEs) is defined as an event not present prior to the initiation of the treatments or any event already present that worsens in either intensity or frequency following exposure to the treatments. AEs occurring more than 3 days after the last day study drug is taken in the study will not be included in the statistical analyses or summaries (except for subjects with adverse events leading to study drug withdrawn). Only treatment-emergent adverse events occurring during the treatment period of the BPS-MR-PAH-202 study will be summarized. Any adverse event starting prior to the first dose of study drug will be excluded from the summary analyses and only presented in the data listings. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Up to 56 months
Measure: Count of Participants; unit: Participants
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 18
Participants | 18

2. Primary Outcome: Number of Treatment Emergent Adverse Events Reported During The Study
Description: A treatment-emergent adverse event (TEAE) is defined as an event not present prior to the initiation of the treatment or any event already present that worsens in either intensity or frequency following exposure to the treatment. AEs occurring more than 3 days after the last day study drug was taken in the study was not included in the statistical analyses or summaries (except for participants with adverse events leading to study drug withdrawn). Only TEAEs that occurred during the treatment period of the BPS-MR-PAH-202 study were summarized. Any adverse event starting prior to the first dose of study drug was excluded from the summary analyses and only presented in the data listings. All efficacy results are descriptive; no statistical analysis was conducted. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Up to 56 months
Measure: Number; unit: TEAEs
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 18
TEAEs | 156

3. Secondary Outcome: Mean Change From Baseline in Six Minutes Walk Distance (6MWD) at End of Study
Description: The area used for the Six Minute Walk Test (6MWT) was pre-measured at a minimum of 30 meters in length and at least 2 to 3 meters in width. There were no turns or significant curves to the 6-minute walk area. The length was marked with gradations to ensure the accurate measurement of the distance walked. The area was well ventilated with air temperature controlled at 20 to 23°C. Intermittent rest periods were allowed if the participant could no longer continue. If the participant needed to rest briefly, he/she could stand or sit and then begin again when rested but the clock continued to run. At the end of 6 minutes, the tester called "stop" while simultaneously stopping the watch and then measured the distance walked. For the purposes of the 6MWT if a participant was assessed at Baseline using oxygen therapy, then all future 6MWT were conducted in the same manner. All efficacy results are descriptive; no statistical analysis was conducted.
Time Frame: Baseline and 56 months
Population: Only participants with both a measurement at baseline and at the given visit are presented.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 11
meters | 10.55 (79.17)

4. Secondary Outcome: Change From Baseline in Borg Dyspnea Score at End of Study
Description: The modified 0-10 category-ratio Borg scale consists of an 11-point scale rating the maximum level of dyspnea experienced during the 6MWT. Scores range from 0 (for the best condition) and 10 (for the worst condition) with nonlinear spacing of verbal descriptors of severity corresponding to specific numbers. The participant chose the number or the verbal descriptor to reflect presumed ratio properties of sensation or symptom intensity. Baseline was defined as the last non-missing evaluation preceding the first dose of study drug in study BPS-MR-PAH-201. Only participants with both a measurement at baseline and at the given visit are presented. All efficacy results are descriptive; no statistical analysis was conducted.
Time Frame: Baseline and 56 months
Population: Only participants with both a measurement at baseline and at the given visit are presented.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 11
scores on a scale | -0.09 (2.84)

5. Secondary Outcome: Number of Participants That Experienced Clinical Worsening During the Study
Description: Number of Participants that experienced Clinical Worsening in the opinion of the Investigator. Clinical Worsening was defined as any of these events following the Baseline visit: Death, Transplantation or atrial septostomy, Clinical deterioration as defined by: Hospitalization as a result of PAH symptoms or Initiation of any new PAH specific therapy (e.g. ERA, PDE-5 inhibitor, prostanoid). All efficacy results are descriptive; no statistical analysis was conducted.
Time Frame: Up to 56 months
Measure: Count of Participants; unit: Participants
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 18
Participants
  Death | 1
  New PAH Therapies | 6
  Transplantation or atrial septostomy | 0
  Hospitalization | 0

6. Secondary Outcome: Number of Participants With a Change in WHO Functional Class
Description: Change from Baseline in participant clinical status was recorded according to the World Health Organization (WHO) Functional Class. A change from lower to higher functional class (i.e. 'III to IV' or 'II to III') was considered as a deterioration. A change from higher to lower functional class (i.e. 'III to II' or 'II to I') was considered as an improvement. All efficacy results are descriptive; no statistical analysis was conducted.
Time Frame: Baseline and 56 months
Measure: Number; unit: Participants
Arm/Group | Beraprost Sodium
Number analyzed (Participants) | 18
Participants
  Improved: Change from Class III to Class II | 1
  No Change in Class | 7
  Deteriorated: Change from Class II to Class III | 4
  Not Reported | 6

ADVERSE EVENTS:
Time Frame: From baseline to 30 days after study treatment discontinuation, up to 56 months.
Arm/Group | Beraprost Sodium
All-Cause Mortality (participants affected / at risk) | 1/18
Serious Adverse Events (participants affected / at risk) | 7/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Beraprost Sodium (N=18)
Right ventricular failure (Cardiac disorders) | 2
Worsening Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Presyncope (Nervous system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Gastroenteritis viral (Infections and infestations) | 1
Syncope (Nervous system disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Bronchitis (Infections and infestations) | 1
Atrial septal defect repair (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Beraprost Sodium (N=18)
Anaemia (Blood and lymphatic system disorders) | 3
Arrhythmia (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 4
Right ventricular heave (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Astigmatism (Eye disorders) | 1
Cataract (Eye disorders) | 1
Eyelid Cyst (Eye disorders) | 1
Myopia (Eye disorders) | 1
Retinal Detachment (Eye disorders) | 1
Retinal Tear (Eye disorders) | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Defaecation urgency (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 1
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Rectal Hemmorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 1
Chest Pain (General disorders) | 1
Fatigue (General disorders) | 2
Generalised oedema (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Biliary Colic (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Hepatitis acute (Hepatobiliary disorders) | 1
Seasonal Allergy (Immune system disorders) | 1
Bronchiolitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 3
Fungal skin infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 6
Urinary Tract Infections (Infections and infestations) | 1
Liver Function Test Abnormal (Investigations) | 1
Platelet Count Decreased (Investigations) | 1
Urine analysis abnormal (Investigations) | 1
Weight increased (Investigations) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Lactose Intolerance (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 5
Headache (Nervous system disorders) | 6
Hypoaesthesia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Restless Leg Syndrome (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 3
Panic Attack (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Worsening pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Skin Irritation (Skin and subcutaneous tissue disorders) | 1
Tooth Extraction (Surgical and medical procedures) | 1
Flushing (Vascular disorders) | 6
Peripheral Coldness (Vascular disorders) | 1
Vasculitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days